CLINICAL TRIAL: NCT05622227
Title: 68Ga-P16-093 PET/CT Imaging in Primary and Recurrent Breast Cancer Patients
Brief Title: 68Ga PET/CT Imaging in Breast Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-BCa093
Record Dates: First submitted 2022-11-14; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-P16-093 and 18F-FDG scan (Experimental): Within 1 week, each patient underwent 68Ga-P16-093 and 18F-FDG PET/CT scan after intravenous administration of 68Ga-P16-093 and 18F-FDG, respectively.
  Interventions: Diagnostic Test: Drug: 68Ga-P16-093

INTERVENTIONS:
Diagnostic Test: Drug: 68Ga-P16-093 — Intravenous injection of 68Ga-P16-093 with the dosage of 1.5-1.8 MBq (0.04-0.05 mCi)/kg. Tracer doses of 68Ga-P16-093 will be used to image lesions of breast cancer by PET/CT.

SUMMARY:
PSMA is highly expressed on the cell surface of the microvasculature of several solid tumors, including breast cancer. This makes it a potentially imaging target for the detection and grading of breast cancer. This pilot study was designed to evaluate the diagnostic performance of 68Ga-P16-093, a novel radiopharmaceutical targeting PSMA, which was compared with 18F-FDG in the same group of breast cancer patients.

DETAILED DESCRIPTION:
PSMA has been confirmed to be over expressed in vascular endothelial cells of various malignant solid tumors, such as breast cancer and renal cancer, which can provide growth advantages for various cancers by cutting the signal molecules involved in angiogenesis. Positron emission tomography (PET) imaging using radiolabeled molecules targeting PSMA can detect a variety of non prostate cancer solid tumors such as breast cancer and glioma. According to previous studies, PSMA can detect primary and metastasis lesions of breast cancer patients, and has a higher uptake value in triple negative breast cancer and HER2 overexpressed patients. The uptake may be related to tumor grade.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients highly suggested by ultrasound or histologically confirmed;
* 68Ga-P16-093 PET/CT and 18F-FDG within two weeks;
* signed written consent.

Exclusion Criteria:

* known allergy against PSMA;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | through study completion, an average of 1 year
  comparing the number of tumor detected by 68Ga-P16-093 and 18F-FDG

SECONDARY OUTCOMES:
standardized uptake value (SUV) of tumor | through study completion, an average of 1 year
  comparing the SUVmax of tumor of different lesions derived from 68Ga-P16-093 AND 18F-FDG

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China